CLINICAL TRIAL: NCT01608880
Title: Effect of Nitroglycerin Ointment on Mastectomy Flap Necrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H12-01161
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Mastectomy Flap Necrosis
MeSH Terms: interventions — polysporin ointment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polysporin Control (Placebo Comparator): Patients in control group will receive polysporin ointment application. Polysporin ointment will be made to look like Nitroglycerin ointment.
  Interventions: Drug: Polysporin ointment
- Nitroglycerin (Active Comparator): Patients in treatment group will receive nitroglycerin ointment application
  Interventions: Drug: nitroglycerin ointment

INTERVENTIONS:
Drug: nitroglycerin ointment — Nitroglycerin ointment will be applied to mastectomy skin flaps at the end of surgery. A maximum of 7.5cm strip of 2% Nitroglycerin ointment will be applied (equivalent to a maximal dose of 45mg)
  Arms: Nitroglycerin
Drug: Polysporin ointment — Polysporin ointment will be applied as the control ointment on the mastectomy flap skin at the end of surgery. A maximum of 7.5cm strip of ointment will be applied to the skin.
  Arms: Polysporin Control

SUMMARY:
Background:

Mastectomy flap necrosis (MFN) is a common complication that affects recovery, reconstructive success and aesthetic outcome. Nitroglycerin (NTG) ointment is a potent topical vasodilator that increases local blood flow by dilating arteries and veins without altering the ratio of pre- to post-capillary resistance. There are no studies that evaluate whether the application of NTG ointment in patients undergoing Skin-sparing mastectomy (SSM) or nipple-sparing mastectomy (NSM) and immediate reconstruction decreases the rate of mastectomy flap necrosis.

Objective:

To evaluate if the post-operative application of NTG ointment improve rates of MFN in patients undergoing SSM or NSM with immediate breast reconstruction compared to patients receiving placebo.

Hypothesis:

In patients undergoing SSM and immediate breast reconstruction there will be a decrease in the rate of MFN in those who receive NTG ointment compared to those who receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo SSM or NSM with immediate alloplastic or autologous breast reconstruction
* Unilateral and bilateral cases (in bilateral cases only the mastectomy performed by the general surgeon will be included. This will avoid the potential effect of absorption of nitroglycerin from one breast to the other)
* Patients older than 21 and less than 65

Exclusion Criteria:

* Patient declining inclusion in the study
* Patient with medical history that precludes the administration of nitroglycerin, i.e. a medical history significant for

  * Acute circulatory failure accompanied by clear hypotension
  * Myocardial insufficiency related to obstruction
  * Use of sildenafil, vardenafil & tadalafil
  * Use of beta-blockers, calcium channel blockers, diuretics or phenothiazides
  * Salicylates (ASA)
  * Alteplase
  * Recent history of MI or cardiac insufficiency
  * Anemia, severe
  * Cerebral hemorrhage or recent head trauma
  * Glaucoma
  * Hepatic function impairment, severe
  * Hyperthyroidism
  * Hypertrophic cardiomyopathy
  * Hypotension
  * Sensitivity to nitrites
* Patient with a history of mantle radiation
* Patient with an allergy to polysporin or any of its ingredients

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mastectomy Flap Necrosis | 1 month post operative

CONTACTS AND LOCATIONS:
Overall Officials: Sheina Macadam, MD, MSc, FRCSC, Principal Investigator — University of British Columbia; Perry Gdalevitch, MD, FRCSC, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Mount Saint Joseph Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia

REFERENCES:
- [Result] Kutun S, Ay AA, Ulucanlar H, Tarcan O, Ay A, Aldan M, Gorkem G, Demir A, Cetin A. Is transdermal nitroglycerin application effective in preventing and healing flap ischaemia after modified radical mastectomy? S Afr J Surg. 2010 Nov;48(4):119-21. PMID 21542401
- [Result] Fan Z, He J. Preventing necrosis of the skin flaps with nitroglycerin after radical resection for breast cancer. J Surg Oncol. 1993 Jul;53(3):210. doi: 10.1002/jso.2930530319. No abstract available. PMID 8331946
- [Result] Rohrich RJ, Cherry GW, Spira M. Enhancement of skin-flap survival using nitroglycerin ointment. Plast Reconstr Surg. 1984 Jun;73(6):943-8. doi: 10.1097/00006534-198406000-00016. PMID 6427801
- [Result] Wong AF, McCulloch LM, Sola A. Treatment of peripheral tissue ischemia with topical nitroglycerin ointment in neonates. J Pediatr. 1992 Dec;121(6):980-3. doi: 10.1016/s0022-3476(05)80356-7. PMID 1447671
- [Result] Jones JT, Stenson MA, Spannagel BD, Robinson DD. Treatment of pressure ulcers with nitropaste. J Am Geriatr Soc. 1997 Jul;45(7):895. doi: 10.1111/j.1532-5415.1997.tb01528.x. No abstract available. PMID 9215351
- [Result] Nelson R. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD003431. doi: 10.1002/14651858.CD003431.pub2. PMID 17054170
- [Result] Fenton C, Wellington K, Easthope SE. 0.4% nitroglycerin ointment : in the treatment of chronic anal fissure pain. Drugs. 2006;66(3):343-9. doi: 10.2165/00003495-200666030-00006. PMID 16526822
- [Result] Rao R, Saint-Cyr M, Ma AM, Bowling M, Hatef DA, Andrews V, Xie XJ, Zogakis T, Rohrich R. Prediction of post-operative necrosis after mastectomy: a pilot study utilizing optical diffusion imaging spectroscopy. World J Surg Oncol. 2009 Nov 25;7:91. doi: 10.1186/1477-7819-7-91. PMID 19939277
- [Result] Losken A, Styblo TM, Schaefer TG, Carlson GW. The use of fluorescein dye as a predictor of mastectomy skin flap viability following autologous tissue reconstruction. Ann Plast Surg. 2008 Jul;61(1):24-9. doi: 10.1097/SAP.0b013e318156621d. PMID 18580145
- [Result] Chun YS, Verma K, Rosen H, Lipsitz SR, Breuing K, Guo L, Golshan M, Grigorian N, Eriksson E. Use of tumescent mastectomy technique as a risk factor for native breast skin flap necrosis following immediate breast reconstruction. Am J Surg. 2011 Feb;201(2):160-5. doi: 10.1016/j.amjsurg.2009.12.011. Epub 2010 Apr 20. PMID 20409522
- [Result] Antony AK, Mehrara BM, McCarthy CM, Zhong T, Kropf N, Disa JJ, Pusic A, Cordeiro PG. Salvage of tissue expander in the setting of mastectomy flap necrosis: a 13-year experience using timed excision with continued expansion. Plast Reconstr Surg. 2009 Aug;124(2):356-363. doi: 10.1097/PRS.0b013e3181aee9a3. PMID 19644248
- [Result] Kroll SS, Ames F, Singletary SE, Schusterman MA. The oncologic risks of skin preservation at mastectomy when combined with immediate reconstruction of the breast. Surg Gynecol Obstet. 1991 Jan;172(1):17-20. PMID 1985335
- [Result] Patani N, Mokbel K. Oncological and aesthetic considerations of skin-sparing mastectomy. Breast Cancer Res Treat. 2008 Oct;111(3):391-403. doi: 10.1007/s10549-007-9801-7. Epub 2007 Oct 28. PMID 17965954
- [Result] Foster RD, Esserman LJ, Anthony JP, Hwang ES, Do H. Skin-sparing mastectomy and immediate breast reconstruction: a prospective cohort study for the treatment of advanced stages of breast carcinoma. Ann Surg Oncol. 2002 Jun;9(5):462-6. doi: 10.1007/BF02557269. PMID 12052757
- [Result] Garwood ER, Moore D, Ewing C, Hwang ES, Alvarado M, Foster RD, Esserman LJ. Total skin-sparing mastectomy: complications and local recurrence rates in 2 cohorts of patients. Ann Surg. 2009 Jan;249(1):26-32. doi: 10.1097/SLA.0b013e31818e41a7. PMID 19106672
- [Result] Sacchini V, Pinotti JA, Barros AC, Luini A, Pluchinotta A, Pinotti M, Boratto MG, Ricci MD, Ruiz CA, Nisida AC, Veronesi P, Petit J, Arnone P, Bassi F, Disa JJ, Garcia-Etienne CA, Borgen PI. Nipple-sparing mastectomy for breast cancer and risk reduction: oncologic or technical problem? J Am Coll Surg. 2006 Nov;203(5):704-14. doi: 10.1016/j.jamcollsurg.2006.07.015. Epub 2006 Sep 11. PMID 17084333
- [Result] Crowe JP, Patrick RJ, Yetman RJ, Djohan R. Nipple-sparing mastectomy update: one hundred forty-nine procedures and clinical outcomes. Arch Surg. 2008 Nov;143(11):1106-10; discussion 1110. doi: 10.1001/archsurg.143.11.1106. PMID 19015470
- [Derived] Gdalevitch P, Brasher P, Macadam S. Reply: Effects of Nitroglycerin Ointment on Mastectomy Flap Necrosis in Immediate Breast Reconstruction: A Randomized Controlled Trial. Plast Reconstr Surg. 2016 Apr;137(4):748e. doi: 10.1097/01.prs.0000481832.83256.5d. No abstract available. PMID 27018703
- [Derived] Gdalevitch P, Van Laeken N, Bahng S, Ho A, Bovill E, Lennox P, Brasher P, Macadam S. Effects of nitroglycerin ointment on mastectomy flap necrosis in immediate breast reconstruction: a randomized controlled trial. Plast Reconstr Surg. 2015 Jun;135(6):1530-1539. doi: 10.1097/PRS.0000000000001237. PMID 26017589